CLINICAL TRIAL: NCT05567497
Title: Evaluating the Perioperative Analgesic Effect of Ultrasound-guided Trigeminal Nerve Block in Adult Patients Undergoing Maxillo-facial Surgery Under General Anesthesia: A Randomized Controlled Study
Brief Title: Ultrasound Guided Trigeminal Nerve Block in Maxillofacial Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trigeminal nerve block
Record Dates: First submitted 2022-09-25; First posted 2022-10-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2022-12

CONDITIONS: Maxillofacial Injuries
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trigeminal Nerve Block (TNB) (Active Comparator): patients will receive general anesthesia followed 5 ml of 0.25% Bupivacaine for TGB under USG after induction of anesthesia (Block Group).
  Interventions: Procedure: trigeminal nerve block
- control (No Intervention): patients will receive general anesthesia only (Control Group).

INTERVENTIONS:
Procedure: trigeminal nerve block — ultrasound guided trigeminal nerve block
  Arms: Trigeminal Nerve Block (TNB)

SUMMARY:
This study aims to evaluate the perioperative analgesic effect of USG Trigeminal Nerve Block in adult patients undergoing maxillofacial surgery. We hypothesized that giving USG-guided TNB in patients undergoing maxilla-facial surgery could reduce the requirements of opioids perioperatively and avoid the side effects of opioids used.

The aim of this double-blind study is to evaluate the effect of USG-guided TNB intra- and post-operatively in terms of pain relief, opioid consumption and adverse effects in patients undergoing such elective surgeries.

DETAILED DESCRIPTION:
Nerve block using various agents has been proposed as a part of the multimodal analgesia to decrease consumption of intravenous opioids and also decrease its complications such as respiratory depression. Recent research has focused on the role of trigeminal nerve blocks (TNB) for management of facial pain . This block was found to be effective in trigeminalneuralgia , palate surgeries and oral and dental surgeries.

Anatomically, the Gasserian ganglion lies in the middle cranial fossa within the Meckel's cave and gives rise to three branches (1) ophthalmic, (2) maxillary, and (3) mandibular which exit from skull through three distinct foramina: the superior orbital fissure, the foramen rotundum, and the foramen ovale. The injection anterior and medial to lateral pterygoid plate into the upper part of pterygopalatine fossa (PPF) will place the injectate in close vicinity to foramen rotundum from where drug migrates into the middle cranial fossa. Since the PPF is extremely vascular, visualizing vascular and soft tissue structures in real time minimize the potential inadvertent complications.

Fluoroscopy-guided blocks have long been considered the gold standard practice in head and neck pain management. Alternatively, computed tomography-guided procedures provide a useful option but expensive and have radiation hazard. Lately, ultrasonography (USG) has been used extensively for perioperative pain relief providing excellent visualization of soft tissue and vasculature with real-time needle placement.

To date, very few published studies had evaluated the value of USG-guided TNB for control of perioperative pain in maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesia (ASA) criteria I/II
* Scheduled for elective unilateral maxillo-facial surgery

Exclusion Criteria:

* Patients with polytrauma and fracture base of skull.
* Patients with known allergy to the study drugs.
* Patients with coagulopathy.
* Patients with infection at puncture site.
* Patients necessitating postoperative ventilation from the start, since it will be difficult to assess respiratory depression and postoperative pain.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
total fentanyl consumption during the intraoperative period. | immediately at the end of the surgery
  the amount of the fentanyl that will be used intraoperatively as analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No